CLINICAL TRIAL: NCT05094518
Title: A Mobile Health Intervention to Increase Uptake of Prenatal Care in Syrian Refugee Population in Turkey
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: HERA Inc (Other)
Collaborators: Medical Rescue Association (MEDAK), Turkey (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: HeraInc
Record Dates: First submitted 2021-09-07; First posted 2021-10-26 (Actual); Last update posted 2021-10-26 (Actual); Status verified 2021-10

CONDITIONS: Prenatal Care; Pregnancy
Keywords: Mobile health; Refugee

STUDY DESIGN:
Intervention Model Description: The intervention group cluster will use the HERA application to receive appointment reminders. The Informed and Non-Informed Control groups will not be using the HERA application.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Reminder (Experimental): Participants will fill the sociodemographic and health history form. Participants will receive reminders in the form of push notifications for prenatal checkup dates automatically generated according to their pregnancy start data or initial check-up appointment for 6 months. Reminders will be sent at the following intervals: 1) 2 weeks before the appointment, 2) 1 day before the appointment, and 3) on the day of appointment. After this date, participants will receive push notifications asking whether they went to the appointment or not weekly for 1 month. This reminder algorithm will be used for each prenatal checkup for a total of four appointments: once in first trimester, once in second trimester and two in third trimester, using the World Health Organization and Turkish Ministry of Health prenatal checkup calendar. At the end of 6 months of follow up period, participants will be contacted via phone call to ask for any remaining appointments or unanswered notifications.
  Interventions: Behavioral: Mobile phone reminders
- Informed Control No Reminder (No Intervention): Participants will fill the sociodemographic and health history form. Their contact information will be gathered. Participants will be contacted at the end of 6 months and will be asked about the number of the prenatal care appointments they have attended during their pregnancy.
- Uninformed Control No Reminder (No Intervention): Participants will fill the sociodemographic and health history form. No contact information will be gathered. The purpose of this arm is to estimate the "true" baseline for the number of visits without any extra attention given by the medical staff.

INTERVENTIONS:
Behavioral: Mobile phone reminders — Appointment reminders in the form of push notifications will be sent through HERA app.
  Arms: Reminder

SUMMARY:
The purpose of this study is to assess the effectiveness of mobile phone based appointment reminder notifications sent through Health Recording App (HERA) in increasing the uptake of 4 World Health Organization recommended prenatal visits among Syrian refugee population.

DETAILED DESCRIPTION:
Background: 12 million Syrians have been forcibly displaced from their homes since the start of Syrian Civil War in 2011. Despite Turkey providing free healthcare services through national insurance to nearly 4 million refugees that it hosts, pregnant Syrian women are less likely to attend prenatal visits and more likely to die during and after labor. An increase in the uptake of prenatal care may improve quality of life through healthy pregnancies and safer labor conditions in this population with double vulnerability.

Mobile phone-based reminders have been shown in randomized controlled trials and systematic reviews to increase the uptake of various services, including prenatal care. Mobile phone penetration is high among Syrian refugees in Turkey and qualitative studies demonstrate that mobile health interventions are acceptable and feasible for Syrian refugees.

Primary objective: To evaluate the impact of mobile phone-based reminders on the uptake of prenatal care among pregnant Syrian refugee women. More specifically, the study assesses the effectiveness of mobile phone-based reminders by measuring the percent increase in the number of prenatal appointments attended by intervention arm participants compared to the control arm participants.

Study design: This is a behavioral intervention study using an un-blinded, parallel groups, randomized controlled study design.

Primary Outcome:

The primary outcome of this study is the number of medical visits, following the initial baseline prenatal care visit, over the 6 month period prior to childbirth.

Secondary outcomes:

Secondary outcomes are based on the Sociodemographic and Health History form. The form gathers information about demographics of the participants (age, education, employment, marital status, number of children) and health history (previous pregnancies, delivery methods, miscarriages, stillborn, chronic conditions and medications. We will further examine these risk factors on the number of medical visits during the study period.

ELIGIBILITY:
Inclusion Criteria:

* Having the status of "Syrian under temporary protection"
* Being in the first trimester of the pregnancy
* Initial prenatal visit
* Age equal or greater than 18 years and less than or equal to 49

Exclusion Criteria:

* Having a citizenship or a status other than "Syrian under temporary protection"
* Not owning a mobile phone
* Being unable to read and write
* Not initial prenatal visit
* Having a chronic disorder or high-risk pregnancy that requires the individual to go to the hospital frequently. Frequently is defined as more than 3 visits post the baseline visit.
* While gestating, those that develop a high-risk pregnancy that requires more than 3 visits post the baseline visit.

Ages: 18 Years to 49 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 162 (Estimated)
Dates: Start 2021-12-01 (Estimated); Primary Completion 2022-12-01 (Estimated); Study Completion 2022-12-01 (Estimated)

PRIMARY OUTCOMES:
Rate of attendance for prenatal care visits | 6 months
  The number of 4 mandatory prenatal care appointments that are attended are presented here.

SECONDARY OUTCOMES:
Sociodemographic and Health information form data | 6 months
  Data about sociodemographic and health information of participants will be presented here.

CONTACTS AND LOCATIONS:
Overall Officials: Aral Surmeli, MD, Principal Investigator — Founder/CEO

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-10-21): https://cdn.clinicaltrials.gov/large-docs/18/NCT05094518/Prot_SAP_000.pdf
  • Informed Consent Form (2021-10-21): https://cdn.clinicaltrials.gov/large-docs/18/NCT05094518/ICF_001.pdf